CLINICAL TRIAL: NCT05782738
Title: A Randomized Clinical Study Comparing Reverse T-stenting and Minimal Protrusion With External Minicrush for Treatment of Complex Coronary Bifurcation (T-REX Trial)
Brief Title: Reverse T-stenting and Minimal Protrusion With External Minicrush for Treatment of Complex Coronary Bifurcation
Acronym: T-REX
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Enrico Cerrato, Interventional Cardiology, San Luigi Gonzaga Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 001-2023
Record Dates: First submitted 2023-03-11; First posted 2023-03-24 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Coronary Disease
Keywords: Reverse TAP; External Minicrush; Coronary bifurcation lesion
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Coronary Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reverse TAP (Active Comparator)
  Interventions: Procedure: Percutaneous Coronary Intervention
- External Minicrush (Active Comparator)
  Interventions: Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Use dedicated two stents technique for treatment of coronary bifurcation stenosis

SUMMARY:
The Reverse T-stenting And Minimal Protrusion (Reverse TAP) is an up-front 2-stent technique that treats complex coronary bifurcation. Compared to crush techniques, it does not require crushing of the side branch stent but only minimal protrusion of the side branch stent before main vessel stenting. Nowadays, no studies compare the Reverse-TAP and the External Minicrush in treating complex coronary bifurcation, so eventually, procedural, clinical and safety differences remain unknown.

DETAILED DESCRIPTION:
According to DEFINITION criteria, PCI of the complex coronary bifurcation with up-front two stent techniques is associated with lower target vessel revascularisation (TVR) than Provisional Stenting. The Double-Kissing Crush stenting (DK-Crush) has been tested with the Culotte and the Classic Crush techniques in the unprotected left main disease (ULMD) and in no-ULMD setting, respectively, showing better clinical outcomes. However, due to its technical complexity and simultaneous improvement of the Classic Crush technique in the External Minicrush, the latter has become the most used technique in the clinical practice in treating complex coronary bifurcation. The DK-Crush technique has never been tested with the External Minicrush, leaving the operators to choose one or the other according to their experience and preferences. The Reverse T-stenting, And Minimal Protrusion (Reverse TAP) is an up-front 2-stent technique that treats complex coronary bifurcation. Compared to crush techniques, it does not require crushing of the side branch stent but only minimal protrusion of the side branch stent before main vessel stenting. Nowadays, studies need to compare the Reverse-TAP and the External Minicrush in treating complex coronary bifurcation, so eventually, procedural, clinical and safety differences remain unknown.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old;
* Patients with an indication of PCI, including Chronic Coronary syndrome (CCS) and Acute Coronary Syndrome (ACS), according to current guidelines recommendations; According to Medina and Definition criteria, patients with at least true and complex coronary lesions involved in coronary bifurcation.

Exclusion Criteria:

* Patients that refused informed consent;
* Patients without valid vascular access that could make unsafe PCI;
* Patients with an expected life of less than one year;
* Patients with scheduled major surgery that required prolonged DAPT interruption;
* Pregnant patients;
* Patients with DAPT contraindications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure (TLF) (Composite of all causes of death, non-fatal TVMI, ischemia-driven target lesion revascularisation (TLR) + Definite or probable ST+ ISR >50% at planned coronary angiography or Coro-TC. | 12-moths
  The investigators check eventually differences in technical and clinical performance between the two techniques through coronary angiography or Coro-TC (centre preferences).

SECONDARY OUTCOMES:
Cardiac death + TVMI + ST | 5-years
  The investigators check mid-term cardiovascular clinical performance between the two techniques.
Cardiac death + TVMI + ST +TLR | 5-years
  The investigators check mid-term cardiovascular clinical performance between the two techniques, including any revascularization of the target lesion site.

OTHER OUTCOMES:
Acute closure of the side branch and periprocedural-MI. | Periprocedural
  The investigators check safety of procedural profile between two techniques.
Intraprocedural ST and periprocedural-MI | Periprocedural
  The investigators check safety of procedural profile between two techniques.
Major bleeding (BARC 3 and 5) | 5-years
  The investigators check safety of hemorrhagic profile between two techniques in consideration of prolonged DAPT.
Technical success | Procedural
  Defined as TIMI flow 3 and < 30% residual stenosis after PCI on target vessel
Procedural success | Periprocedural
  Defined as technical success with no in-hospital major adverse
Cross-over between groups | Periprocedural
  Possibility to switching between two techniques for technical reasons
Timing of rewiring | Periprocedural
  Measure of the time spending in a crucial phase of the two techniques
Number of guide wire used | Periprocedural
  Number of coronary guidewires to perform the assigned technique.
Amount of contrast medium used | Periprocedural
  Total contrast medium used to perform the PCI with the technique assigned
Procedural time | Periprocedural
  Total time used to perform the PCI
Fluoroscopic time | Periprocedural
  Total fluoroscopic time spending to perform the PCI
X-rays exposition | Periprocedural
  Total operators x-rays exposition during the PCI

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Piedimonte, MD, Principal Investigator — Ospedale degli Infermi di Rivoli (TO)
Locations (5):
- Italy (5):
  - Ciriè Hospital, Cirié, Tori O
  - Ospedale Santa Croce, Moncalieri, Torino
  - Azienda ospedaliera Santi Antonio e Biagio e Cesare Arrigo, Alessandria
  - L'Azienda Ospedaliera (AO) S. Croce e Carle, Cuneo
  - Interventional Unit, San Luigi Gonzaga University Hospital, Orbassano, and Rivoli Hospital, Turin, Italy, Turin

IPD SHARING:
Plan to Share IPD: No